CLINICAL TRIAL: NCT05004987
Title: Depression Treatment and Aβ Dynamics: A Study of Alzheimer's Disease Risk (ABD Study)
Brief Title: Aβ Dynamics in LLMD
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21-00535
Record Dates: First submitted 2021-08-12; First posted 2021-08-13 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Alzheimer Disease; Major Depressive Disorder
MeSH Terms: conditions — Alzheimer Disease; Depressive Disorder, Major | interventions — Escitalopram

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Both the study staff and the subjects will be blind to the study assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Escitalopram (ESC) (Active Comparator)
  Interventions: Drug: Escitalopram Oxalate
- Placebo (PBO) (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Escitalopram Oxalate — The daily dose of ESC/PBO will be 10 mg for the first 2 weeks, then increase to 20 mg as tolerated, with an option to reduce back to 10 mg if necessary.
  Other Names: Lexapro; ESC
  Arms: Escitalopram (ESC)
Drug: Placebo — Daily dose of placebo will mimic that of ESC.
  Other Names: PBO
  Arms: Placebo (PBO)

SUMMARY:
This study will examine the biological factors that may modulate the relationship between depression and the development of Alzheimer's disease (AD). Since the direction of causation between depression and the biological factors associated with AD is unknown, the only way to understand cause and associated risk is to treat the depressive symptoms and examine the effects on AD biomarkers. The study involves an FDA-approved treatment for major depressive disorder. It will compare the SSRI antidepressant escitalopram with placebo. The hypothesis is that a reduction in depressive symptoms will be associated with a normalization of CSF AD biomarkers as well as peripheral inflammatory markers. This research would contribute to fundamental knowledge about potentially modifiable risks of Alzheimer's disease (AD).

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects, age 60+ years inclusive, at the time of signing the informed consent.
2. Meeting Structured Clinical Interview (SCID-5-RV) for DSM-5 criteria for Major depressive disorder.
3. Montgomery-Åsberg Depression Rating Scale (MADRS) ≥18.
4. Have results of a physical examination, neurological examination, vitals, and EKG within normal limits at screening.
5. Cognitively unimpaired at screening visit as defined by Mini-Mental State Examination (MMSE) >27.
6. Clinical Dementia Rating Scale (CDR) Global of 0*.
7. A score of 85 or greater on the RBANS delayed memory index score.
8. Fluent in English, because some of the instruments used in this study have not been translated and validated in other languages, and are able to read at a 6th grade level or equivalent, as determined by the PI.
9. Medically stable with no significant cerebrovascular, neurological, or systemic disease expected to interfere with the study.
10. Adequate auditory acuity and normal-to-corrected vision.
11. Willing to undergo brain MRI, urine drug screen and blood sampling for routine laboratory testing, lumbar puncture, APOE genotyping and plasma drug levels.
12. Only individuals with normal or non-clinically significant abnormalities on routine laboratory tests, will be included.

    * If study partner is not available, the CDR will be skipped.

Exclusion Criteria:

1. History of brain tumor, MRI evidence of brain damage or brain disease including significant trauma, hydrocephalus, seizures, or confluent (or more extensive) white matter hyperintensities.
2. Mental retardation, or other serious neurological disorder (e.g. Parkinson's disease or other movement disorders).
3. Subjects with a Fazekas scale >2.
4. Significant history of alcoholism or drug abuse in the past 2 years. Fulfilling SCID-5-RV/DSM-5 criteria for current or past diagnosis of any psychiatric disorder (e.g., schizophrenia, bipolar disorder, or any psychotic disorder) other than recurrent MDD or anxiety disorders (e.g., panic disorder, agoraphobia, etc.).
5. A current significant risk for suicidality based on the Columbia-Suicide-Severity Rating Scale (C-SSRS).
6. Insulin dependent diabetes.
7. Evidence of clinically relevant or unstable cardiac, pulmonary, endocrine or hematological conditions.
8. Any prosthetic devices (e.g., pacemaker or surgical clips) that constitutes a hazard for MRI imaging.
9. Positive urine drug screen for illicit drugs.
10. History of poor tolerance to, poor response to, or ongoing treatment with escitalopram.
11. If taking antidepressants, currently taking fluoxetine, due to the length of time required to washout.
12. Treatment with following medications will not be permitted. In some cases, medications will be allowed if medically prescribed and dose regimen stable. Note: Some medications (e.g., amphetamines, opiates) may appear on the routine urine drug test in the screening period but can be allowed as per protocol.

    * For subjects taking prescribed psychoactive medications and supplements (i.e., opioids, amphetamines, amphetamine-like substances, and cannabinoids), must be on a stable dose for 1 month prior to randomization.
    * Anti-Parkinsonian medications (carbidopa/levodopa, amantadine, bromocriptine, pergolide, selegiline).
    * Cholinesterase inhibitors and memantine
    * Continuous aspirin (any dosage) use which can affect platelet function is prohibited. Exception: If participant is on low dose aspirin for prophylaxis and is willing to temporarily discontinue prior to research blood draw (i.e., 2 days before).
    * Continuous use of other medications which are also known to affect platelet function, including nonsteroidal anti-inflammatory drugs (NSAIDs), anti-histamines. Exception: If participant is taking medication continuously and is willing to temporarily discontinue prior to research blood draw (i.e., 2 days before)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-02-04 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-01-29 (Estimated)

PRIMARY OUTCOMES:
Change in Cerebrospinal Fluid (CSF) Aβ40 Biomarker Levels | Baseline, Week 8
Change in Cerebrospinal Fluid (CSF) Aβ42 Biomarker Levels | Baseline, Week 8
Change in Vascular Dysfunction (VD) Biomarker Levels | Baseline, Week 8
Change in Scores on Montgomery-Asberg Depression Ration Scale (MADRS) | Baseline, Week 8
  MADRS consists of 10 items evaluating core symptoms of depression (e.g, apparent sadness, reported sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thought, and suicidal thoughts). Each symptom is rated on a 0-6 scale (0=no abnormality, 6=severe). The total score ranges from 0 to 60; the higher the score, the more severe the symptoms.

OTHER OUTCOMES:
Change in Plasma Aβ Biomarker Levels | Baseline, Week 8
Change in Cerebrospinal Fluid (CSF) P-tau Biomarker Levels | Baseline, Week 8
Change in Cerebrospinal Fluid (CSF) T-tau Biomarker Levels | Baseline, Week 8

CONTACTS AND LOCATIONS:
Overall Officials: Nunzio Pomara, MD, Principal Investigator — NYU Langone Health
Locations (2):
- United States (2):
  - NYU Langone Health, New York, New York
  - Nathan S. Kline Institute for Psychiatric Research, Orangeburg, New York

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be shared upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will have access to the data upon reasonable request. Requests should be directed to nunzio.pomara@nki.rfmh.org. To gain access, data requestors will need to sign a data access agreement.